CLINICAL TRIAL: NCT06949332
Title: Electromyographic Investigation of the Instant Effect of Rocabado Exercise Approaches on Masseter Muscle Activity
Brief Title: Investigation of the Instant Effect of Rocabado Exercise
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Emre Serdar Atalay, doctoral faculty member, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: 2024-456
Record Dates: First submitted 2025-04-08; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Electromyography; Exercise; Temporomandibular Joint Disc Displacement
Keywords: rocabado exercise; Temporomandibular Joint Disc; electromyography; superficial electromyography; emg; exercise
MeSH Terms: conditions — Motor Activity | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy sedentary group: Healthy, sedentary individuals aged 18-40. No history of bruxism or increased masticatory muscle tone.
  Protocol:
  EMG: Masseter muscle activity during 6 Rocabado exercises. Tragus-to-Wall Distance: Cervical/upper thoracic posture. Maximum active mouth opening. Lateral Mandibular Mobility: Sideways jaw movement. Oral parafunctional habits. Neck pain and disability level.
  Interventions: Device: electromyography

INTERVENTIONS:
Device: electromyography — In this study, surface Electromyography (EMG) was employed to assess the electrical activity of the masseter muscles. Surface EMG is a physiological measurement technique that allows for the recording of electrical potentials generated by muscle fiber depolarization through non-invasive electrodes placed on the skin. This method is widely accepted for objectively determining muscle activation levels and timing, enabling the quantitative analysis of changes in masseter muscle activity during the performance of various Rocabado exercises in this study. The validity and reliability of the EMG device utilized (Noraxon USA Inc., Scottsdale, AZ, USA) have been established in the literature.

SUMMARY:
The temporomandibular joint (TMJ) or jaw joint is a bilateral hinge joint formed by the fusion of the temporal bone and mandible, which provides complex movements necessary for basic functions such as eating, swallowing, speaking and yawning. This joint, which can perform rotation and translation movements, functions with the coordinated work of the masticatory muscles (masseter, temporalis, pterygoideus medialis and lateralis, digastricus). The masseter muscle in particular plays an important role in closing the jaw and generating chewing force.

Rocabado exercises are a special exercise program that requires the active participation of the patient to restore the normal movement of the TMJ, reduce pain, maintain body balance and correct postural disorders. This program includes six different exercises: tongue relaxation position, shoulder retraction, head position stabilization, chin tuck, TMJ rotation control and rhythmic stabilization technique.

There are a limited number of studies on the effectiveness of Rocabado exercises in the literature and there is no study specifically examining the effects of these exercises on the masseter muscle. Therefore, this study will investigate the effects of Rocabado exercises on masseter muscle activity in sedentary individuals. The findings may provide a new perspective in the physiotherapy processes of individuals with masseter muscle problems and may contribute to the selection of appropriate exercises to increase the activation of this muscle by determining which Rocabado exercise activates the masseter muscle more.

DETAILED DESCRIPTION:
This study aims to investigate the effect of different Rocabado exercises on masseter muscle activity in healthy, sedentary individuals. The study will be conducted at the Faculty of Physiotherapy and Rehabilitation, Health Sciences University Gülhane, Ankara, Türkiye.

Participants and Recruitment

A total of 35 healthy, sedentary individuals aged between 18 and 40 years will be recruited for this study. Participants will be included based on the following criteria:

Age between 18 and 40 years. No engagement in any regular sports activities (sedentary lifestyle). Voluntary participation in the study.

Individuals will be excluded if they have:

A history of teeth grinding or bruxism. Clinical signs of increased muscle tone in the masticatory muscles upon physical examination by a physiotherapist.

A masseter pressure pain threshold measurement below a predetermined cutoff point, as assessed by an algometer (Baseline, USA). This criterion is included to ensure participants do not have underlying muscle sensitivity that could influence EMG readings.

Recruitment will be conducted through online announcements on social media platforms and messaging applications. Interested individuals who meet the inclusion criteria will be selected for participation. Prior to their involvement, all participants will provide written informed consent after receiving a detailed explanation of the study's purpose, procedures, potential risks, and benefits, both orally and in written form. The study schedule will be determined, and willing participants will be invited to the research facility. A physiotherapist will assess the participants for any signs of increased masticatory muscle tone and will include them in the study based on this assessment.

Data Collection

The following data will be collected from each participant:

Demographic and Health Data: Information such as name, age, education level, and relevant medical history will be recorded.

Masseter Muscle Activity Assessment via Electromyography (EMG): Surface EMG (Noraxon USA Inc., Scottsdale, AZ, USA) will be used to measure the electrical activity of the masseter muscles. Participants will be tested individually in a quiet environment. They will be seated comfortably, and their demographic information (height, weight, etc.) will be recorded in the EMG device. Before the test, participants will be instructed on how to perform each of the six Rocabado exercises. The physiotherapist will demonstrate each exercise. The exercises will be performed in a randomized order for each participant to minimize any potential order effects on the EMG data. Non-invasive surface electrodes will be placed bilaterally over the masseter muscles in a manner that does not cause discomfort . EMG data will be recorded during the performance of each exercise.

The Noraxon USA Inc. surface EMG device, along with its electrodes and signal processing units , is a validated and reliable instrument for assessing muscle activation. Surface EMG detects muscle activity through non-invasive electrodes applied to the skin surface . During each exercise, the real-time EMG signal will be monitored on the device screen and recorded for subsequent analysis .

Tragus-to-Wall Distance Measurement: This measurement will be taken to assess the participants' cervical and upper thoracic posture . Participants will stand with their feet shoulder-width apart, heels, buttocks, and shoulders against a wall. They will be instructed to maintain a "good posture," looking straight ahead, and to hold this position during the measurement. The distance between the tragus of the ear and the wall will be measured using a ruler.

Maximum Active Mouth Opening (MAMO) Measurement: Participants will be asked to open their mouths as wide as possible without causing pain. The distance between the upper and lower incisal edges will be measured in millimeters using a ruler. Three trials will be performed, and the average value will be recorded .

Lateral Mandibular Mobility Measurement: This measurement assesses the distance of lateral movement between the upper and lower central incisors. The mandible should move symmetrically in a specific plane during lateral excursions, with movement typically being equal on both sides and less than 8 mm.

Oral Habits Checklist (OBC): The "Oral Behaviour Checklist (OBC)," a 21-item questionnaire, will be administered to identify parafunctional habits such as day and night teeth clenching, teeth grinding, nail biting, lip or cheek biting, pen biting, and gum chewing, which are known to play a significant role in the pathogenesis of Temporomandibular Disorders (TMD).

Neck Disability Index (NDI): The Turkish version of the Neck Disability Index, a 10-item questionnaire developed by Dr. Howard Vernon and validated for Turkish population by Telci et al. , will be used to assess the participants' neck pain levels and the impact of neck pain on their daily activities. Each question has a score ranging from 0 to 5, with a maximum total score of 50. If participants do not drive or work, those specific questions will be excluded from the scoring.

Rocabado Exercise Protocol

Participants will perform each of the following six Rocabado exercises with 6 repetitions each, as described below:

Tongue Relaxation Position: With teeth apart and lips closed, the anterior one-third of the tongue rests on the palate, without touching the teeth. Diaphragmatic breathing is performed through the nose.

Shoulder Retraction: The shoulders are simultaneously moved downwards and backwards, bringing the shoulder blades together.

Cervical Retraction (Head Positioning): With hands clasped behind the neck to stabilize it, the head is gently moved forward (chin tuck) and then returned to the starting position (distraction movement).

Chin Tucks (Jaw Movement): The chin is moved towards the neck and then away, maintaining a straight horizontal movement.

Controlled TMJ Rotation: In the tongue relaxation position, the index finger is placed on the TMJ while controlled mouth opening and closing movements are performed. Lateral deviation of the jaw is avoided. Participants will be encouraged to perform this exercise in front of a mirror to ensure proper control and to learn controlled chewing patterns.

Rhythmic Stabilization Technique: In the tongue resting position, the index finger is placed on the chin to stabilize the jaw. The participant is asked to apply a slight resistance while performing small opening, closing, and lateral deviation movements of the TMJ.

Statistical Analysis Demographic data obtained from the participants will be presented using descriptive statistics (e.g., mean, standard deviation, frequency, percentage). The normality of the data for the outcome measures (EMG activity during each exercise, tragus-to-wall distance, MAMO, lateral mandibular mobility) will be assessed using the One-Sample Kolmogorov-Smirnov test. If the data are normally distributed, a one-way repeated measures analysis of variance (ANOVA) will be used to compare the masseter muscle activity during the six different Rocabado exercises. In case of non-normal distribution, the non-parametric Friedman test will be used for the same comparison. The level of statistical significance will be set at p < 0.05 for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years.
* No engagement in any regular sports activities (sedentary lifestyle).
* Voluntary participation in the study.

Exclusion Criteria:

* A history of teeth grinding or bruxism.
* Clinical signs of increased muscle tone in the masticatory muscles upon physical examination by a physiotherapist.
* A masseter pressure pain threshold measurement below a predetermined cutoff point, as assessed by an algometer (Baseline, USA). This criterion is included to ensure participants do not have underlying muscle sensitivity that could influence EMG readings.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy sedentary individuals
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Masseter Muscle Activition | immediate effect during exercise
  Masseter muscle activation, refers to the summation of electrical potentials generated by the motor units of the masseter muscle fibers upon stimulation by motor nerves. This physiological process enables muscle contraction and consequently, the elevation of the mandible (upward movement of the jaw) and the execution of masticatory function. The intensity and duration of activation vary according to the applied force and the phase of the chewing cycle, and it can be non-invasively measured using methods such as surface EMG.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | before exercise
  his is a self-report questionnaire consisting of 10 items that assess the impact of neck pain on a person's daily activities and their perceived level of disability. It covers areas such as pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Higher scores indicate a greater level of disability due to neck pain.
Oral Habits Checklist | before exercise
  This is a self-report questionnaire comprising 21 items designed to evaluate the frequency and nature of various parafunctional oral behaviors that the individual has engaged in over the past month. These behaviors include teeth grinding and clenching (during sleep and wakefulness), nail biting, lip or cheek biting, tongue thrusting, gum chewing, and others. The checklist aims to quantify the occurrence of these habits, which are often associated with temporomandibular disorders (TMD).

OTHER OUTCOMES:
demographic information | before exercise
  Age, weight, height and dominant side information were taken and entered into the noraxon system. These demographic data will be collected to describe the general characteristics of the participant group and to assess possible influencing factors. As mentioned in the statistical analysis section, these demographic data will be presented as descriptive statistics.
Tragus Wall Distance Measurement | before exercise
  It will be measured for the evaluation of neck and upper back posture. Tragus wall distance measurement will be used to assess spinal mobility. Participants will be asked to stand with feet shoulder width apart, heels, hips and shoulders against the wall. Participants will then be asked to "stand in a good posture, look straight ahead and maintain this position until the measurement is made". The distance between the tragus and the wall at the participant's ear level will be measured
Maximum Active Mouth Opening Measurement | before exercise
  For the measurement of maximum active mouth opening, the participant will be asked to open the mouth as wide as possible without pain. The distance between the upper and lower incisors will be measured in millimeters with a ruler. After 3 trials, the average will be taken
Measurement of lateral mobility of the jaw | before exercise
  It is the measurement of the lateral shift distance between the anterior middle teeth. The mandible should move symmetrically in a certain plane during movement. Lateralization movements should be equal on both sides and less than 8mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Health Sciences Faculty, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Is core stability training effective in temporomandibular disorder? A randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/37924356/
- See also: Electromyographic analysis of the masseter and buccinator muscles with the pro-fono facial exerciser use in bruxers — https://pubmed.ncbi.nlm.nih.gov/16541843/
- See also: Masseter Muscle Thickness And Elasticity in Bruxism After Exercise Treatment: A Comparison Trial — https://pubmed.ncbi.nlm.nih.gov/36057478/